CLINICAL TRIAL: NCT01904136
Title: A Phase I/II Clinical Trial of NK Cells Administration to Prevent Disease Relapse for Patient With High-Risk Myeloid Malignancies Undergoing Haploidentical Stem-Cell Transplantation
Brief Title: Natural Killer Cells Before and After Donor Stem Cell Transplant in Treating Patients With Acute Myeloid Leukemia, Myelodysplastic Syndrome, or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0708; NCI-2013-02183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01 - 5P01; RP110553 05-07-04832; 05-07-04832; 2012-0708 (Other: M D Anderson Cancer Center); P01CA049639 (NIH)
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia With Gene Mutations; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; de Novo Myelodysplastic Syndrome; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Stem Cell Transplantation; Bone Marrow Transplantation; Blood Specimen Collection; Cyclophosphamide; fludarabine; Melphalan; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (NK cells, allogeneic stem cell transplant) (Experimental): MYELOABLATIVE CONDITIONING REGIMEN: Patients receive high-dose melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and NK cells IV over 30 minutes on day -2 or -1.
  NON-MYELOABLATIVE CONDITIONING REGIMEN: Patients receive melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and receive NK cells IV over 30 minutes on day -2 or -1.
  TRANSPLANT: Patients undergo allogeneic PBSC or bone marrow transplant on day 0.
  POST-TRANSPLANT CYCLOPHOSPHAMIDE AND GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days 3 and 4, tacrolimus IV beginning on day 5 for 2 weeks and then PO for approximately 4 months, and mycophenolate mofetil PO TID beginning on day 5 for approximately 6-7 months.
  NK CELLS: Patients receive NK cells IV over 30 minutes on days 7 and 28-90.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Mycophenolate Mofetil; Biological: Natural Killer Cell Therapy; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSC or bone marrow transplant
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Procedure: Bone Marrow Transplantation — Undergo allogeneic PBSC or bone marrow transplant
  Other Names: Blood and Bone Marrow Transplant; BMT; Bone Marrow Grafting; Bone Marrow Transplant; Marrow Transplantation
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given PO
  Other Names: CellCept; MMF
Biological: Natural Killer Cell Therapy — Given IV
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSC or bone marrow transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation

SUMMARY:
This phase I/II studies the side effects and best dose of natural killer cells before and after donor stem cell transplant and to see how well they work in treating patients with acute myeloid leukemia, myelodysplastic syndrome, or chronic myelogenous leukemia. Giving chemotherapy with or without total body irradiation before a donor peripheral blood stem cell or bone marrow transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells and natural killer cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate safety, tolerability and identify the maximum tolerated dose (MTD) of expanded natural killer (NK) cells to be used in patients with myeloid malignancies undergoing a haploidentical stem-cell transplant.

SECONDARY OBJECTIVES:

I. To determine survival of NK cells in vivo post-transplant. II. To determine the function of NK cells post-transplant and compare with a retrospective control treated with no NK cells.

III. To estimate the proportion of patients with engraftment/graft failure. IV. To estimate the non-relapse mortality (NRM) at day 100 post-transplant. V. To estimate the cumulative incidence of grade III-IV aGVHD (acute graft-versus-host disease) at day 100.

VI. To assess the rate of chronic graft-versus-host disease (GVHD) within the first year post transplantation.

VII. To assess immune reconstitution post-transplant. VIII. To assess disease response, disease-free survival (DFS) and overall survival (OS) after transplantation.

IX. To perform a retrospective comparison of patients treated on the study with NK cells will be performed with a Center for International Blood and Marrow Transplant Research (CIBMTR) control of similar patients who did not receive NK cells.

OUTLINE: This is a phase I, dose-escalation study of NK cells followed by a phase II study. Patients are assigned to 1 of 2 conditioning regimens.

MYELOABLATIVE CONDITIONING REGIMEN: Patients receive high-dose melphalan intravenously (IV) over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo total-body irradiation (TBI) on day -3, and NK cells IV over 30 minutes on day -2 or -1.

NON-MYELOABLATIVE CONDITIONING REGIMEN: Patients receive melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and receive NK cells IV over 30 minutes on day -2 or -1.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell (PBSC) or bone marrow transplant on day 0.

POST-TRANSPLANT CYCLOPHOSPHAMIDE AND GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days 3 and 4, tacrolimus IV beginning on day 5 for 2 weeks and then orally (PO) for approximately 4 months, and mycophenolate mofetil PO thrice daily (TID) beginning on day 5 for approximately 6-7 months.

NK CELLS: Patients receive NK cells IV over 30 minutes on days 7 and 28-90.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for pediatric patients will be determined in conjunction with an MD Anderson Cancer Center (MDACC) pediatrician; patients age 2-17 years old may be enrolled after at least 4 adults (ages 18-65 years old) have been treated without toxicity
* Patient with no matched related donor who has a related haploidentical donor identified (=< 7/8 allele match at the A, B, C, DR loci) who is willing to undergo a bone marrow harvest and an NK cell collection approximately 2 weeks of the recipient's admission for transplant; the donor must be 16 years of age or older and weigh at least 110 pounds
* Patients with one of the following diseases: acute myeloid leukemia (AML): a. first complete remission with high-risk features defined as: (i) greater than 1 cycle of induction therapy required to achieve remission; (ii) preceding myelodysplastic syndrome (MDS); (iii) presence of FLT3 mutations or internal tandem duplication or other mutations associated with poor-risk AML (e.g. DNMT3A, TET2); (iv) French-American-British Classification (FAB) M6 or M7 classification; (v) adverse cytogenetics: -5, deletion (del) 5q, -7, del7q, abnormalities involving 3q, 9q, 11q, 20q, 21q, 17, +8 or complex karyotype (> 3 abnormalities); (vi) treatment-related AML, or b. second or greater remission; patients beyond second remission have to be in complete remission (CR) at transplant to be eligible, or c. primary induction failure with partial response to therapy who achieve adequate cytoreduction
* Patients with myelodysplastic syndromes (MDS): a. de novo MDS with intermediate or high-risk International Prognostic Scoring System (IPSS) scores; patients with intermediate-1 features should have failed to respond to hypomethylating agent therapy, or b. patients with treatment-related MDS
* Chronic myeloid leukemia (CML): a. failed to achieve cytogenetic remission or have cytogenetic relapse after treatment with at least 2 tyrosine kinase inhibitors, or b. accelerated phase or blast phase at any time
* Performance score of at least 70% by Karnofsky or 0 to 1 by Eastern Cooperative Oncology Group (ECOG) (age >= 12 years), or Lansky Play-performance scale of at least 70% or greater (age < 12 years)
* Serum creatinine clearance equal or more than 50 ml/min (calculated with Cockcroft-Gault formula)
* Bilirubin equal or less than 1.5 mg/dl except for Gilbert's disease
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) equal or less than 200 IU/ml for adults
* Conjugated (direct) bilirubin less than 2 x upper limit of normal
* Left ventricular ejection fraction equal or greater than 40%
* Diffusing capacity of the lung for carbon monoxide (DLCO) equal or greater than 50% predicted corrected for hemoglobin; for children =< 7 years of age who are unable to perform pulmonary function tests (PFT), oxygen saturation >= 92% on room air by pulse oximetry
* Patient or patient's legal representative, parent(s) or guardian should provide written informed consent; assent of a minor if participant's age is at least seven and less than eighteen years

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive; active hepatitis B or C
* Uncontrolled infections; principal investigator (PI) is the final arbiter of this criterion
* Liver cirrhosis
* Central nervous system (CNS) involvement within 3 months
* Positive pregnancy test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization
* Inability to comply with medical therapy or follow-up

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samer Srour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ciurea SO, Kongtim P, Soebbing D, Trikha P, Behbehani G, Rondon G, Olson A, Bashir Q, Gulbis AM, Indreshpal K, Rezvani K, Shpall EJ, Bassett R, Cao K, Martin AS, Devine S, Horowitz M, Pasquini M, Lee DA, Champlin RE. Decrease post-transplant relapse using donor-derived expanded NK-cells. Leukemia. 2022 Jan;36(1):155-164. doi: 10.1038/s41375-021-01349-4. Epub 2021 Jul 26. PMID 34312462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at MD Anderson Cancer Center from April 2014 until June 2019.
Pre-assignment Details: Total number of participants registered in MDACC was 54, which 27 participants were Donors (Signed consent but not involved in results outcome and no Adverse events were collected) and 27 were Recipients (Treated with donor NK cells).
Groups:
- Phase I: NK Cell Dose Level 1_10^4; Phase I: NK Cell Dose Level 2_10^5; Phase I: NK Cell Dose Level 3_10^6; Phase I: NK Cell Dose Level 4_ 10^7; Phase I: NK Cell Dose Level 5_3x10^7; Phase I: NK Cell Dose Level 6_10^8: MYELOABLATIVE CONDITIONING REGIMEN: Patients receive high-dose melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and NK cells IV over 30 minutes on day -2 or -1.
  NON-MYELOABLATIVE CONDITIONING REGIMEN: Patients receive melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and receive NK cells IV over 30 minutes on day -2 or -1.
  TRANSPLANT: Patients undergo allogeneic PBSC or bone marrow transplant on day 0.
  POST-TRANSPLANT CYCLOPHOSPHAMIDE AND GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days 3 and 4, tacrolimus IV beginning on day 5 for 2 weeks and then PO for approximately 4 months, and mycophenolate mofetil PO TID beginning on day 5 for approximately 6-7 months.
  NK CELLS: Patients receive NK cells IV over 30 minutes on days 7 and 28-90.
  Cohort 1: 1xE4 Cohort 2: 1xE5 Cohort 3: 1xE6 Cohort 4: 1xE7 Cohort 5: 3xE7 Cohort 6: 1xE8
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic PBSC or BMT
  Cyclophosphamide: Given IV Fludarabine: Given IV Laboratory Biomarker Analysis: Correlative studies Melphalan: Given IV Mycophenolate Mofetil: Given PO Natural Killer Cell Therapy: Given IV Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSC or BMT Tacrolimus: Given IV and PO Total-Body Irradiation: Undergo TBI
- Phase II: NK Cell Dose Level 5_3x10^7; Phase II: NK Cell Dose Level 6_10^8: MYELOABLATIVE CONDITIONING REGIMEN: Patients receive high-dose melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and NK cells IV over 30 minutes on day -2 or -1.
  NON-MYELOABLATIVE CONDITIONING REGIMEN: Patients receive melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and receive NK cells IV over 30 minutes on day -2 or -1.
  TRANSPLANT: Patients undergo allogeneic PBSC or bone marrow transplant on day 0.
  POST-TRANSPLANT CYCLOPHOSPHAMIDE AND GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days 3 and 4, tacrolimus IV beginning on day 5 for 2 weeks and then PO for approximately 4 months, and mycophenolate mofetil PO TID beginning on day 5 for approximately 6-7 months.
  NK CELLS: Patients receive NK cells IV over 30 minutes on days 7 and 28-90.
  Cohort 5: 3xE7 Cohort 6: 1xE8
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic PBSC or BMT
  Cyclophosphamide: Given IV Fludarabine: Given IV Laboratory Biomarker Analysis: Correlative studies Melphalan: Given IV Mycophenolate Mofetil: Given PO Natural Killer Cell Therapy: Given IV Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSC or BMT Tacrolimus: Given IV and PO Total-Body Irradiation: Undergo TBI
- Donor: KIR mismatched haplo donors, KIR mismatched cord blood donors or HLA matched related donors.
Period: Overall Study
Arm/Group | Phase I: NK Cell Dose Level 1_10^4 | Phase I: NK Cell Dose Level 2_10^5 | Phase I: NK Cell Dose Level 3_10^6 | Phase I: NK Cell Dose Level 4_ 10^7 | Phase I: NK Cell Dose Level 5_3x10^7 | Phase I: NK Cell Dose Level 6_10^8 | Phase II: NK Cell Dose Level 5_3x10^7 | Phase II: NK Cell Dose Level 6_10^8 | Donor
Started | 1 | 2 | 3 | 3 | 2 | 3 | 3 | 10 | 27
Completed | 1 | 2 | 3 | 3 | 2 | 2 | 3 | 10 | 27
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twenty seven donor participants only signed consents and were not part of the results outcome and Adverse events were not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: NK Cell Dose Level 1_10^4 | Phase I: NK Cell Dose Level 2_10^5 | Phase I: NK Cell Dose Level 3_10^6 | Phase I: NK Cell Dose Level 4_ 10^7 | Phase I: NK Cell Dose Level 5_3x10^7 | Phase I: NK Cell Dose Level 6_10^8 | Phase II: NK Cell Dose Level 5_3x10^7 | Phase II: NK Cell Dose Level 6_10^8 | Donor | Total
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 3 | 3 | 10 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 4
  Between 18 and 65 years | 1 | 2 | 3 | 2 | 2 | 3 | 3 | 10 | 24 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 1 | 3 | 1 | 5 | 11 | 25
  Male | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 5 | 16 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 6
  Not Hispanic or Latino | 1 | 2 | 2 | 3 | 2 | 2 | 3 | 9 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3 | 3 | 2 | 2 | 3 | 10 | 27 | 53
  Iran | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Number of participants that experienced dose limiting toxicities.
Time Frame: Up to day 70 post-transplant
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: NK Cell Dose Level 5_3x10^7; Phase II: NK Cell Dose Level 6_10^8: MYELOABLATIVE CONDITIONING REGIMEN: Patients receive high-dose melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and NK cells IV over 30 minutes on day -2 or -1.
  NON-MYELOABLATIVE CONDITIONING REGIMEN: Patients receive melphalan IV over 30 minutes on day -7, fludarabine IV over 1 hour on days -7 to -4, undergo TBI on day -3, and receive NK cells IV over 30 minutes on day -2 or -1.
  TRANSPLANT: Patients undergo allogeneic PBSC or bone marrow transplant on day 0.
  POST-TRANSPLANT CYCLOPHOSPHAMIDE AND GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days 3 and 4, tacrolimus IV beginning on day 5 for 2 weeks and then PO for approximately 4 months, and mycophenolate mofetil PO TID beginning on day 5 for approximately 6-7 months.
  NK CELLS: Patients receive NK cells IV over 30 minutes on days 7 and 28-90.
  Cohort 5: 3xE7 Cohort 6: 1xE8
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic PBSC or BMT Cyclophosphamide: Given IV Fludarabine: Given IV Laboratory Biomarker Analysis: Correlative studies Melphalan: Given IV Mycophenolate Mofetil: Given PO Natural Killer
Arm/Group | Phase I: NK Cell Dose Level 1_10^4 | Phase I: NK Cell Dose Level 2_10^5 | Phase I: NK Cell Dose Level 3_10^6 | Phase I: NK Cell Dose Level 4_ 10^7 | Phase I: NK Cell Dose Level 5_3x10^7 | Phase I: NK Cell Dose Level 6_10^8 | Phase II: NK Cell Dose Level 5_3x10^7 | Phase II: NK Cell Dose Level 6_10^8 | Donor
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 2 | 3 | 10 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: 100-day Treatment Related Mortality
Description: Number of participants who died within 100 days post-transplant.
Time Frame: Up to 100 days post-transplant
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: NK Cell Dose Level 1_10^4 | Phase I: NK Cell Dose Level 2_10^5 | Phase I: NK Cell Dose Level 3_10^6 | Phase I: NK Cell Dose Level 4_ 10^7 | Phase I: NK Cell Dose Level 5_3x10^7 | Phase I: NK Cell Dose Level 6_10^8 | Phase II: NK Cell Dose Level 5_3x10^7 | Phase II: NK Cell Dose Level 6_10^8 | Donor
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 2 | 3 | 10 | 0
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0

3. Secondary Outcome: Overall Survival
Description: Number of participants with overall survival after 2 years.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: NK Cell Dose Level 1_10^4 | Phase I: NK Cell Dose Level 2_10^5 | Phase I: NK Cell Dose Level 3_10^6 | Phase I: NK Cell Dose Level 4_ 10^7 | Phase I: NK Cell Dose Level 5_3x10^7 | Phase I: NK Cell Dose Level 6_10^8 | Phase II: NK Cell Dose Level 5_3x10^7 | Phase II: NK Cell Dose Level 6_10^8 | Donor
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 2 | 3 | 10 | 0
Participants | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 5 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Description: Twenty seven donor participants only signed consents and were not part of the results outcome and Adverse events were not collected.
Arm/Group | Phase I: NK Cell Dose Level 1_10^4 | Phase I: NK Cell Dose Level 2_10^5 | Phase I: NK Cell Dose Level 3_10^6 | Phase I: NK Cell Dose Level 4_ 10^7 | Phase I: NK Cell Dose Level 5_3x10^7 | Phase I: NK Cell Dose Level 6_10^8 | Phase II: NK Cell Dose Level 5_3x10^7 | Phase II: NK Cell Dose Level 6_10^8 | Donor
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/2 | 1/3 | 0/3 | 0/2 | 0/2 | 1/3 | 5/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/2 | 3/3 | 0/3 | 0/2 | 0/2 | 2/3 | 6/10 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 3/3 | 3/3 | 2/2 | 2/2 | 3/3 | 10/10 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: NK Cell Dose Level 1_10^4 (N=1) | Phase I: NK Cell Dose Level 2_10^5 (N=2) | Phase I: NK Cell Dose Level 3_10^6 (N=3) | Phase I: NK Cell Dose Level 4_ 10^7 (N=3) | Phase I: NK Cell Dose Level 5_3x10^7 (N=2) | Phase I: NK Cell Dose Level 6_10^8 (N=2) | Phase II: NK Cell Dose Level 5_3x10^7 (N=3) | Phase II: NK Cell Dose Level 6_10^8 (N=10) | Donor (N=0)
Secondary graft failure (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral Infections (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial Infections (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
GI GvHD (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Delayed engraftment (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Liver GvHD (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CNS hemorrahge due to DSA/PLT Refractory (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: NK Cell Dose Level 1_10^4 (N=1) | Phase I: NK Cell Dose Level 2_10^5 (N=2) | Phase I: NK Cell Dose Level 3_10^6 (N=3) | Phase I: NK Cell Dose Level 4_ 10^7 (N=3) | Phase I: NK Cell Dose Level 5_3x10^7 (N=2) | Phase I: NK Cell Dose Level 6_10^8 (N=2) | Phase II: NK Cell Dose Level 5_3x10^7 (N=3) | Phase II: NK Cell Dose Level 6_10^8 (N=10) | Donor (N=0)
Bacterial Infections (Infections and infestations) | 1 | 1 | 3 | 2 | 2 | 1 | 2 | 5 | 0
Flu like syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Neutropenic fevers (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 0 | 2 | 2 | 10 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 2 | 2 | 3 | 10 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 3 | 2 | 2 | 3 | 10 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 5 | 0
Viral Infections (Infections and infestations) | 0 | 1 | 3 | 2 | 2 | 1 | 3 | 10 | 0
Fevers (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0
Fluid overload (General disorders) | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 7 | 0
Skin GvHD (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 4 | 0
GI GvHD (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 0
Elevated bilirubin (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Fungal Infections (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Liver GvHD (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Upper GI GvHD (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 5 | 0
Hemorrhagic Cystitis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Mucositis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 7 | 0
BK virus associated hemorrhagic cystitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 5 | 0
Elevated transminitis (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0
Neutropenic enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytoxan induced Hemorrhagic Cystitis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT01904136/Prot_SAP_000.pdf